CLINICAL TRIAL: NCT00345943
Title: An fMRI Study of Self-regulation in Adolescents With Bulimia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rachel Marsh, Research Scientist, New York State Psychiatric Institute
Other Study IDs: #5606R/6679R; R01MH090062 (NIH); DDTR M2-MBB
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Eating Disorders
Keywords: Eating Disorders; Bulimia Nervosa; Bulimia; fMRI; Magnetic Resonance Imaging
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Bulimia | interventions — Diffusion Tensor Imaging; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adolescents with Bulimia Nervosa or subclinical BN: Adolescents with Bulimia Nervosa or subclinical Bulimia Nervosa
  Interventions: Other: MRI; Behavioral: Neuropsychological Testing
- Healthy control adolescents: Healthy control adolescents
  Interventions: Other: MRI; Behavioral: Neuropsychological Testing

INTERVENTIONS:
Other: MRI — Magnetic Resonance Imaging scans
  Other Names: GE 3T scanner; Anatomical Images, DTI, and MRS
Behavioral: Neuropsychological Testing — Neuropsychological tests
  Other Names: Wechsler Abbreviated Scale of Intelligence (WASI); Continuous Performance Task; Stroop Word-Color Interference; Weather Prediction Task

SUMMARY:
The aim of this project is to use both multimodal MRI and behavioral measures to investigate how changes in frontostriatal neural systems contribute to the development and persistence of Bulimia Nervosa (BN). Findings from this study will have wide-ranging importance for our understanding of the development and treatment of BN.

DETAILED DESCRIPTION:
Patients with Bulimia Nervosa (BN) have difficulty regulating impulsive behaviors as suggested by their binge-eating and purging, as well as the high incidence of drug abuse and shoplifting in this population. Understanding dysfunction in the frontostriatal circuitry that mediates self-regulatory control processes will aid development of new therapeutics for the impulsivity associated with BN. We are conducting a longitudinal study to better understand the development and persistence of BN.

Participation in this study includes 4 sections: Neuropsychological Tests, Diagnostic interviews, Pregnancy Test, and MRI scan. All efforts are made to coordinate procedures into one day, and they require between 4 and 5 hours of the participant's time. The option of splitting participation into two study days is also offered for participants who find it more convenient. Participants are compensated with $100 in the form of a check, which is mailed to their home address. Participants will be invited back for follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Current or prior DSM IV diagnosis of Bulimia Nervosa or Sub-threshold Bulimia Nervosa (those who meet all DSM-IV criteria for BN, but engage in subjective binge-eating episodes and binge/purge at a frequency of at least once per week for 3 months, whereas meeting full DSM-IV criteria for BN requires binge eating and purging twice per week for 3 months)
* Major Depression
* For control adolescents, no current or past history of an eating disorder

Exclusion Criteria:

* Ferromagnetic implants (e.g., pacemaker)
* Metal braces or retainers
* IQ less than 80
* Any other current major Axis I disorder, other than major depressive disorder (MDD)
* History of concussion, seizure disorder, or other neurological illness
* Claustrophobia
* Pregnant

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents (ages 12-17 years) with bulimia nervosa and age, gender, and weight-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2004-10; Primary Completion 2016-09 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Marsh, PhD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute at Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Berner LA, Wang Z, Stefan M, Lee S, Huo Z, Cyr M, Marsh R. Subcortical Shape Abnormalities in Bulimia Nervosa. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Dec;4(12):1070-1079. doi: 10.1016/j.bpsc.2018.12.011. Epub 2019 Jan 4. PMID 30846367
- [Derived] Cyr M, Wang Z, Tau GZ, Zhao G, Friedl E, Stefan M, Terranova K, Marsh R. Reward-Based Spatial Learning in Teens With Bulimia Nervosa. J Am Acad Child Adolesc Psychiatry. 2016 Nov;55(11):962-971.e3. doi: 10.1016/j.jaac.2016.07.778. Epub 2016 Sep 8. PMID 27806864
- [Derived] Marsh R, Maia TV, Peterson BS. Functional disturbances within frontostriatal circuits across multiple childhood psychopathologies. Am J Psychiatry. 2009 Jun;166(6):664-74. doi: 10.1176/appi.ajp.2009.08091354. Epub 2009 May 15. PMID 19448188

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adolescents With Bulimia Nervosa or Subclinical BN | Healthy Control Adolescents
Started | 38 | 33
Completed | 33 | 28
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents With Bulimia Nervosa or Subclinical BN | Healthy Control Adolescents | Total
Number analyzed (Participants) | 33 | 28 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (1.5) | 16.2 (2.1) | 16.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 22 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 28 | 18 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 28 | 61
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.1 (2.8) | 21.4 (3.5) | 21.8 (3.1)
Wechsler Abbreviated Intelligence Scale (WASI) [Mean (Standard Deviation); unit: units on a scale] — This estimates Full Scale IQ with excellent reliability and validity for ages 6-90. The measure is comprised of 4-subtests: block design task, vocabulary task, matrix reasoning test and similarities test. A composite score is calculated by summing the scores on the 4 subtests. Standard score ranges:
  Superior: >130; Very High: 120-129; Bright normal: 110-119; Average: 90-109; Low Average: 80-89; Borderline Mental Functioning: 70-79
  units on a scale | 105.5 (16.1) | 104.9 (11.4) | 105.2 (13.9)
Illness duration [Mean (Standard Deviation); unit: months] — Population: This clinical measure was only administered to the Adolescents with Bulimia Nervosa or subclinical BN group
  months
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 26.0 (19.9) |  | 26.0 (19.9)
Eating Disorder Examination - objective binge eating episodes (past 28 days) [Mean (Standard Deviation); unit: Number of episodes] — Population: This clinical measure was only administered to the Adolescents with Bulimia Nervosa or subclinical BN group
  Number of episodes
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 13.8 (17.8) |  | 13.8 (17.8)
Eating Disorder Examination - subjective binge eating episodes (past 28 days) [Mean (Standard Deviation); unit: Number of episodes] — Population: This clinical measure was only administered to the Adolescents with Bulimia Nervosa or subclinical BN group
  Number of episodes
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 18.3 (24.3) |  | 18.3 (24.3)
Eating Disorder Examination - self-induced vomiting episodes (past 28 days) [Mean (Standard Deviation); unit: Number of episodes] — Population: This clinical measure was only administered to the Adolescents with Bulimia Nervosa or subclinical BN group
  Number of episodes
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 32.9 (28.7) |  | 32.9 (28.7)
Eating Disorder Examination - loss of control episodes (past 28 days) [Mean (Standard Deviation); unit: Number of episodes] — Population: This clinical measure was only administered to the Adolescents with Bulimia Nervosa or subclinical BN group
  Number of episodes
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 25.2 (20.1) |  | 25.2 (20.1)
Comorbid Major Depressive Disorder [Number; unit: participants] — Population: Any lifetime Axis I disorder (including Major Depressive Disorder) was exclusionary for the Healthy control group
  participants
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 14 |  | 14
Comorbid Anxiety Disorders [Number; unit: participants] — Population: Any lifetime Axis I disorders (including Anxiety disorders) was exclusionary for the Healthy Control group
  participants
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 7 |  | 7
Psychotropic Medication Use [Number; unit: participants] — Population: Psychotropic medication use was exclusionary for the Healthy Control group
  participants
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 9 |  | 9
Prior Anorexia Nervosa (%) [Count of Participants; unit: Participants] — Population: Any lifetime Axis I disorders (including Anorexia Nervosa) was exclusionary for the Healthy Control group
  Participants
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 5 |  | 5
Inpatient Treatment [Number; unit: participants] — Population: Ongoing psychiatric treatment was exclusionary for the Healthy control group
  participants
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 13 |  | 13
Outpatient Treatment [Number; unit: participants] — Population: Ongoing psychiatric treatment was exclusionary for the Healthy control group
  participants
    number analyzed (Participants) | 33 | 0 | 33
    (all) | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Imaging Scans
Description: This study will use magnetic resonance imaging (MRI) to assess the structure (cortical thickness) of neural circuit regions involved in Bulimia Nervosa (BN).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Adolescents With Bulimia Nervosa or Subclinical BN | Healthy Control Adolescents
Number analyzed (Participants) | 33 | 28
mm | 2.98 (0.22) | 2.96 (0.22)
Statistical Analysis 1: Comparison: Adolescents With Bulimia Nervosa or Subclinical BN vs Healthy Control Adolescents; Growth curve models examined the following: group (BN versus HC) differences in cortical thickness (CT) at baseline; group differences in the rate of change in CT over time; and the persistence of group differences in CT over time; Test type: Other; p = .03, Mixed Models Analysis; Growth curve models with between-within degrees of freedom and a random effect for the intercept and fixed effects for predictors; Mean Difference (Net) = -0.10, Standard Error of Mean 0.04 — BN versus HC group effect
Statistical Analysis 2: Comparison: Adolescents With Bulimia Nervosa or Subclinical BN vs Healthy Control Adolescents; Growth curve models examined the following: group (BN versus HC) differences in conflict-related BOLD signal at baseline; group differences in the rate of change in conflict-related BOLD signal over time; and the persistence of group differences in conflict-related BOLD signal over time; Test type: Other; p < .05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = 0.053, 95% CI 2-sided [-0.04 to 0.15], Standard Error of Mean 0.047

2. Secondary Outcome: Conners Continuous Performance Test-II (CPT-II)
Description: The Conners Continuous Performance Test-II (CPT-II) is a standardized measure of attention and impulsivity. The following variables (T-scores) were used:
  Omissions: the number of times the participant failed to respond to a target. High T-score indicates a worse outcome.
  Commissions: the number of times the participant responded but no target was presented. High T-score indicates a worse outcome.
  Hit Reaction Time: time between the presentation of the stimulus and participant's response. A fast reaction time (low T-score) and high commission errors points to difficulties with impulsivity. A slow reaction time (high T-score) with high commission and omission errors, indicates inattention in general.
  Hit Reaction Time Standard Error: levels of inconsistency in response speed. High T-score indicates a worse outcome.
  Detectability: discrimination for target and nontarget. High T-score indicates a worse outcome.
  Population mean (standard deviation) = 50 (10)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Adolescents With Bulimia Nervosa or Subclinical BN | Healthy Control Adolescents
Number analyzed (Participants) | 30 | 23
T-scores
  Omissions | 49.52 (12.48) | 53.24 (16.50)
  Commissions | 53.31 (8.25) | 50.20 (12.30)
  Hit Reaction Time | 39.71 (7.33) | 45.57 (13.41)
  Hit Reaction Time Standard Error | 45.81 (9.38) | 49.23 (11.06)
  Detectability | 54.18 (6.47) | 50.98 (10.50)

3. Secondary Outcome: Stroop Word-Color Interference
Description: The Stroop Word-Color Interference Test is a neuropsychological test assessing the ability to inhibit cognitive interference.
  The test contains three parts: word page (the names of colors printed in black ink), color page (rows of X's printed in colored ink) and word-color page (the words from the first page are printed in the colors from the second page; however, the word meanings and ink colors are mismatched).The subject's task is to look at each sheet and move down the columns, reading words or naming the ink colors as quickly as possible, within a given time limit (45 seconds). Three scores, as well as an interference score, are generated using the number of items completed on each page, with higher scores reflecting better performance and less interference on reading ability. Scores range 0-100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescents With Bulimia Nervosa or Subclinical BN | Healthy Control Adolescents
Number analyzed (Participants) | 33 | 28
score on a scale | 22.1 (6) | 21.5 (5)

4. Secondary Outcome: Weather Prediction Task
Description: The Weather Prediction Task is a measure of probabilistic learning using experimental analysis of weather prediction. In this task, participants try to predict either "rain" or "shine" based on the presentation of cards whose cue-outcome associations vary probabilistically. Accuracy score (i.e. percentage of correct response) was used in our analyses. A higher score indicates better outcome. Values range 0-100%, with 50% being chance level.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of correct response
Arm/Group | Adolescents With Bulimia Nervosa or Subclinical BN | Healthy Control Adolescents
Number analyzed (Participants) | 19 | 20
percentage of correct response | 54.9 (11.5) | 51.4 (10.4)

ADVERSE EVENTS:
Time Frame: 5 years (Year 1-5)
Arm/Group | Adolescents With Bulimia Nervosa or Subclinical BN | Healthy Control Adolescents
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/33
Other Adverse Events (participants affected / at risk) | 0/38 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No